CLINICAL TRIAL: NCT06527092
Title: The Effect of Virtual Reality on Pain, Anxiety And Fear During Venipuncture in Children Aged 6-12 Years: A Randomised Controlled Trial
Brief Title: The Effect of VR on Pain, Anxiety And Fear During Venipuncture in Children
Acronym: VR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Dilek Zengin, Asst. Prof., Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 22-7T/31
Record Dates: First submitted 2024-07-23; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Pain, Acute; Anxiety; Fear
Keywords: Venipuncture; Non-pharmacological; Pain; Children; Nursing
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain | interventions — Gastric Balloon

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual reality (Experimental): The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale-Condition (CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) before the procedure. The child was fitted with virtual reality goggles and a video of the child's choice was shown. One of the videos was a video of visiting animals in the zoo, while the other video was an aquarium video containing colorful fish and creatures under the sea. The zoo visit video is 3 minutes 51 seconds and the aquarium visit video is 11 minutes 55 seconds. Two minutes after the child started watching the video, peripheral catheter insertion was started. During the procedure, the same nurse, who was independent of the study, assessed the child with the Child Anxiety Scale-Condition(CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the child's crying (how many seconds it lasted).
  Interventions: Device: Virtual Reality
- Bubbles (Experimental): The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale-Condition(CAS-D), Child Fear Scale and Visual Analogue Scale (VAS) before the procedure. The child was given a colourful, lighted bubble gun. Two minutes after the child used the coloured-light bubble gun, peripheral catheter insertion was started. During the procedure, the same nurse, who was independent from the study, assessed the child with the Child Anxiety Scale-Condition (CAS-D), Child Fear Scale and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the child's crying (how many seconds it lasted).
  Interventions: Device: Bubbles
- Control (No Intervention): The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale- Condition (CAS-D), Child Fear Scale and Visual Analogue Scale (VAS) before the procedure. Peripheral catheter insertion was started. Distraction techniques such as asking questions and talking were used during the procedure. During the procedure, the same nurse, who was independent from the study, evaluated with the Child Anxiety Scale- Condition (CAS-D), Child Fear Scale and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the crying status of the child (how many seconds it lasted).

INTERVENTIONS:
Device: Virtual Reality — VR is an interactive, multidimensional, computer-simulated environment accessed through a head-mounted device that blocks the view of the real world. This environment is projected in front of the user's eyes through sophisticated head-mounted displays, including a wide field of view and motion tracking systems
  Arms: Virtual reality
Device: Bubbles — A colorful light bubble gun was used for bubble therapy, which is one of the distraction methods.
  Arms: Bubbles

SUMMARY:
The use of non-pharmacological applications such as virtual reality,and bubbles are recommended in intravenous interventions. There are very few studies evaluating the effect of non-pharmacological applications in intravenous localization. This study was planned as a randomized controlled trial. The effects of virtual reality and bubble application on pain, fear, anxiety, procedure time and crying time in intravenous insertion were evaluated. Children (105) aged 6-12 years who were treated in a children's hospital and underwent intravenous placement were randomized to virtual reality, bubbles, and control groups. Distraction techniques such as asking questions and talking were used with the children in the control group. Study data were collected using the Child Anxiety Scale-Conditioning (CAS-D), Child Fear Scale, and Visual Analogue Scales (VAS).

DETAILED DESCRIPTION:
The use of non-pharmacological applications such as virtual reality, and bubbles are recommended in intravenous interventions. There are very few studies evaluating the effect of non-pharmacological applications in intravenous localization. This study was planned as a randomized controlled trial. The effects of virtual reality and bubble application on pain, fear, anxiety, procedure time, and crying time in intravenous insertion were evaluated. Children (105) aged 6-12 years who were treated in a children's hospital and underwent intravenous placement were randomized to virtual reality, bubbles, and control groups. Distraction techniques such as asking questions and talking were used with the children in the control group. Study data were collected using the Child Anxiety Scale-Conditioning (CAS-D), Child Fear Scale, and Visual Analogue Scales (VAS).

Virtual reality: The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale-Condition (CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) before the procedure. The child was fitted with virtual reality goggles and a video of the child's choice was shown. One of the videos was a video of visiting animals in the zoo, while the other video was an aquarium video containing colorful fish and creatures under the sea. The zoo visit video is 3 minutes 51 seconds and the aquarium visit video is 11 minutes 55 seconds. Two minutes after the child started watching the video, peripheral catheter insertion was started. During the procedure, the same nurse, who was independent of the study, assessed the child with the Child Anxiety Scale-Condition(CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the child's crying (how many seconds it lasted)

Bubbles: The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale-Condition(CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) before the procedure. The child was given a colorful, lighted bubble gun. Two minutes after the child used the colored-light bubble gun, peripheral catheter insertion was started. During the procedure, the same nurse, who was independent of the study, assessed the child with the Child Anxiety Scale-Condition (CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the child's crying (how many seconds it lasted).

Control: The child was given a comfortable position. A nurse independent from the study assessed the child with the Child Anxiety Scale- Condition (CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) before the procedure. Peripheral catheter insertion was started. Distraction techniques such as asking questions and talking were used during the procedure. During the procedure, the same nurse, who was independent of the study, evaluated with the Child Anxiety Scale- Condition (CAS-D), Child Fear Scale, and Visual Analogue Scale (VAS) and recorded the duration of the procedure and the crying status of the child (how many seconds it lasted).

ELIGIBILITY:
Inclusion Criteria:

- The child was treated at the Ege University Medical Faculty Children's Hospital, Between the ages of 6 and 12, Peripheral catheter insertion Both parents and themselves speak and understand Turkish, and It was determined as volunteering to participate in the study.

Exclusion Criteria:

Children under 6 years of age or over 12 years of age Children treated with analgesics Sedated children

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Procedurel Pain | Six month
  Visual Analogue Scale (VAS): Recommended for use in children aged 7 years and over. The child is asked to mark the level of pain felt on a 10 cm ruler in the range from '0 - no pain' to '10 - most severe pain'. The scale can be used either horizontally or vertically.
Anxiety | Six month
  Child Anxiety Scale-Condition (CAS-D):The CAS-D is shaped like a thermometer with a bulb at the bottom and horizontal lines at intervals going upwards. The score can range from 0 to 10. Turkish validity and reliability have been performed.
Fear | Six month
  Child Fear Scale:The scale is used to measure the fear level of the child. It is a 0-4 scale consisting of five drawn facial expressions ranging from neutral expression (0=no fear) to frightened face (4=severe fear). Turkish validity and reliability have been performed.

SECONDARY OUTCOMES:
duration of crying | Six month
  Follow-up form: Children's crying time will be monitored through this form.

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Zengin, Principal Investigator — Ege University Faculty of Nursing
Locations (1):
- Ege University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No